CLINICAL TRIAL: NCT06551766
Title: The Application of Photosensitive Hydrogel in Intranasal Endoscopic Dacryocystorhinostomy for the Anastomosis of Lacrimal Cyst Flap and Nasal Mucoperiosteal Flap
Brief Title: The Application of Photosensitive Hydrogel in Intranasal Endoscopic Dacryocystorhinostomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023017
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Chronic Dacryocystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photosensitive hydrogel (Experimental): The photosensitive hydrogel is composed of tetra-armed poly(ethylene glycol) (4aPEGNB)and methacrylate-modified hyaluronic acid (HAMA).The hydrogel can be rapidly photocured under light induction at 395nm.
  Interventions: Device: Photosensitive hydrogel
- Suture fixation (Active Comparator): The suture is fixed with 6-0 absorbable thread.
  Interventions: Device: 6-0 absorbable stitches

INTERVENTIONS:
Device: Photosensitive hydrogel — In the photosensitive hydrogel group, the anastomosis of the lacrimal cyst mucosal flap and the nasal mucoperiosteal flap was achieved by photosensitive hydrogel.
  Arms: Photosensitive hydrogel
Device: 6-0 absorbable stitches — In the suture fixation group, the anastomosis of the lacrimal cyst mucosal flap and the nasal mucoperiosteal flap was achieved by two stitches using 6-0 absorbable wire.
  Arms: Suture fixation

SUMMARY:
To study the effect of Photosensitive hydrogel used for suture free anastomosis of lacrimal cyst and nasal mucoperiosteal flap in endoscopic nasal dacryocystostomy, and evaluate its adhesion to lacrimal cyst and nasal mucoperiosteal flap, promoting wound healing, forming a good anastomosis, preventing postoperative anastomosis and shortening operation time. Twenty patients with chronic dacryocystitis were randomly divided into photosensitive hydrogel group and suture group.Symptoms and nasal endoscopy were followed up 2, 6, and 12 weeks after surgery for both groups. And also adverse events were recorded at each follow-up.

DETAILED DESCRIPTION:
After endoscopic dacryocystonasal anastomosis, granulation and/or cicatricial adhesion are the main reasons for surgical failure. How to achieve the ideal fit between the lacrimal sac flap and the nasal mucoperiosteal flap and avoid the proliferation of granulation and cicatricial adhesion is very important for the success of the operation. In this study, "photocoupling reaction" technology was used to achieve seamless integration and strong adhesion of photosensitive hydrogel materials to the wound, and the photohydrogel was applied to suture free adhesion and wound repair of the lacrimal cyst mucosal flap and nasal mucosal flap in endoscopic nasal Dacryocystostomy (En-DCR), and its feasibility, safety and effectiveness were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this clinical study and sign the informed consent;
2. Gender is not limited, age 18-75 years old;
3. The patient had symptoms and signs of chronic dacryocystitis, and the results of lacrimal passage irrigation suggested that the lower rush and return or upper rush and lower return, accompanied by mucous or purulent discharge reflux;
4. Lacrimal duct angiography suggests nasolacrimal duct obstruction without lacrimal canaliculi and/or duct obstruction.

Exclusion Criteria:

1. Age < 18 or > 75 years old;
2. Previous history of dacryocystonasal anastomosis;
3. Abnormal coagulation function;
4. Tumors of lacrimal passage, especially in patients with papilloma or malignant tumors;
5. in the acute dacryocystitis attack stage;
6. obvious scar constitution;
7. Complicated with serious nasal diseases, such as severe allergic rhinitis, chronic rhinosinusitis and nasal polyps, acute suppurative rhinosinusitis, severe atrophic rhinitis, and severe deviation of nasal septum;
8. Have serious heart, liver, kidney, lung and other basic diseases, can not tolerate general anesthesia;
9. Distance from the hospital, postoperative review is not convenient;
10. Participated in other clinical trials within the last 3 months;
11. Any medical history that the investigator determines may interfere with the test results or increase the patient's risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Anastomotic opening rate | 6 weeks after surgery
  The opening of the anastomosis was observed by nasal endoscopy.

SECONDARY OUTCOMES:
Remission rate of tearing symptoms | 2, 6 and 12 weeks after surgery
  The remission of tearing symptoms was assessed by VAS scale

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
We will publish the data in the form of a paper, and other researchers can obtain the required information with the permission of the principal investigator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year
Access Criteria: Other researchers can obtain the required information with the permission of the principal investigator.

DOCUMENTS (1):
  • Study Protocol (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT06551766/Prot_000.pdf